CLINICAL TRIAL: NCT02370797
Title: Lumpectomy Followed by Intraoperative Electron Radiation Therapy (IOERT) as a Single Full Dose Partial Breast Irradiation for Early Stage, Node Negative, Invasive Breast Cancer
Brief Title: Node Negative, Invasive Breast Cancer Single Fraction IOERT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACI-1450-IOERTSFX
Record Dates: First submitted 2015-02-03; First posted 2015-02-25 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: IOERT; Radiation; Single fraction; Lumpectomy; Radiation therapy; Avera
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- Single Fraction IOeRT (Experimental): A single dose of 21 Gy calculated such that the 90% isodose line encompasses the posterior of the tumor bed will be administered.
  Interventions: Radiation: Single Fraction IOeRT

INTERVENTIONS:
Radiation: Single Fraction IOeRT — A single dose of 21 Gy calculated such that the 90% isodose line encompasses the posterior of the tumor bed will be administered.
  Other Names: Intra-Operative electron radiation therapy

SUMMARY:
The purpose of this study is to determine if lumpectomy followed by Intraoperative Electron Radiation Therapy (IOeRT) as a single, full dose partial breast irradiation will have as good or better results in preventing recurrence of local breast cancer, cosmetic appearance and early and late side effects.

DETAILED DESCRIPTION:
See points VIII inclusion/exclusion criteria

Operation:

* Lumpectomy, steninal node biopsy
* IOeRT

After Surgery:

* Meet with a medical oncologist and discuss if chemotherapy and/or hormone therapy is recommended as part of your treatment course. In some cases, pathology results may indicate the need for removal of additional lymph nodes. The doctor will review pathology and discuss if additional surgery is required.
* Chemotherapy (if indicated)
* Hormone therapy (if indicated)

Follow-Up

* Visits will be completed with the surgeon, radiation oncologist and research staff as the protocol indicates.
* Assessements of acute toxicity according to CTC-toxicity scoring system
* Assessments of late toxicity according to LENT-SOMA scoring systems
* Assessment of cosmetic outcome according to scoring system and photo documentation in standardized positions.

ELIGIBILITY:
Inclusion Criteria:

* Patient agrees to breast conservation therapy (segmental resection, partial mastectomy, and radiation therapy) as the treatment for their breast cancer
* Patient agrees to evaluation of the axilla with sentinel lymph node biopsy
* Post-menopausal women age > 60, defined as women who have experienced no menstrual period in the past 12 months.
* BRCA1 and 2 gene mutation negative, if tested. [genetic testing is NOT required based upon personal or family history]
* Unifocal (unicentric), invasive ductal carcinoma or favorable sub-types (mucinous, tubular, colloid) < 2.0 cm in diameter, primary T-stage of T1 (AJCC criteria)
* Grade 1, 2 acceptable
* Associated LCIS is allowed
* Estrogen receptor (ER) status of positive
* Negative margins at ink on gross pathologic examination
* Patient is node-negative, defined as N0 (i-) or N0 (i+)
* Patient must be deemed functionally and mentally competent to understand and sign the informed consent

Exclusion Criteria:

* Prior breast malignancy or other malignancy if metastatic, or with expected survival of < 5 years
* Immuno-compromised status
* Pregnancy
* Women with an active connective tissue disorder (i.e. scleroderma, lupus and others)
* Breast cancer that involves the skin or chest wall, locally advanced breast cancer
* Pure DCIS, all grades
* Invasive lobular carcinoma
* Evidence of lymphovascular invasion (LVI)
* Invasive carcinoma with extensive intraductal component (EIC)
* Neoadjuvant chemotherapy indicated
* Patients with 1 or more positive lymph node determined during surgery with sentinel node and/or axillary dissection
* Not eligible for breast conserving management, i.e., prior whole breast radiation therapy
* Estrogen receptor negative
* Her2 positive
* Grade 3

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2029-02 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are free of breast cancer. | 10 years
  Patients will be followed by standard of care breast imaging along with appointments with breast surgeon, radiation oncologist and medical oncologist if indicated.

SECONDARY OUTCOMES:
Local recurrance rate with acute toxicity and cosmetic evaluations | 10 years
  AEs and Lent Soma will be assessed for acute toxicity. We will use a 20% toxicity cutoff, the protocol would be stopped if 2/10 were determined to have developed significant toxicities, grade 3 or greater, at the first 6-month follow-up visit. 2/10 patients at 6-months follow-up, 4/20 patients at 1-year follow-up, 6/30 at 18-months follow-up, 8/40 at 24-months follow-up, 10/50 at 30-months follow-up, 12/60 at 36-months follow-up, 14/70 at 42-months follow-up, 16/80 at 48-months follow-up, 18/90 at 54-months and 20/100 at 60-months follow-up.
  Cosmetic evaluations will be completed by the patient and radiation oncologist an via breast exams, questionnaires and breast photo documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Arneson, MD, Principal Investigator — Avera Cancer Insitute
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States